CLINICAL TRIAL: NCT01785680
Title: Conducting Research on Moderate Acute Malnutrition in Humanitarian Emergencies Integrated Management of MAM and SAM in Sierra Leone With Ready to Use Theraputic Foods (RUTF)
Brief Title: Moderate Acute Malnutrition (MAM) and Severe Acute Malnutrition (SAM) in Sierra Leone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201211096; U01GH000647-01 (NIH)
Record Dates: First submitted 2013-01-29; First posted 2013-02-07 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Malnutrition
Keywords: MAM; SAM
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Current protocol (Active Comparator): These treatment arm is the standard care for moderate malnutrition. This includes a fortified cereal supplement treatment until the child reaches MUAC of above 12.5. Currently, MAM and SAM are treated separately, overseen by different agencies. Breastfeeding is often overlooked.
  Interventions: Other: Current protocol
- Integrated Protocol (Experimental): Integrated protocol for treatment of children with MAM and SAM in humanitarian emergencies has the potential to result in a more streamlined, cost-effective program, higher recovery, and higher program coverage, allowing easier access to malnourished children, thus curing more children of malnutrition and preventing its lifelong effects.
  Interventions: Other: Integrated Protocol

INTERVENTIONS:
Other: Integrated Protocol — Implement an integrated protocol in Sierra Leone for the management of MAM and non-complicated SAM that uses a single anthropometric indicator as well as the same food but in different doses to treat the continuum of malnutrition. MAM children will be given 75 g/kg/day of RUTF whereas SAM will be given 175 gr/kg/day of RUTF until MUAC>12.5 cm is reached. Then child will be given LNS, a bed net, albendazole, zinc, referral for immunizations compliant with current WHO recommendations, oral rehydration salts to give if the child has more than three loose watery stools in 24 hours, and asked to return for follow-up in 1, 3 and 6 months. Caretakers will be instructed to seek medical care sooner if the child has fever, poor appetite or signs of an acute illness.
  Arms: Integrated Protocol
Other: Current protocol — Current protocol for treating MAM in emergencies is supplemental food distribution, often providing a fortified blended food (FBF) that requires cooking. This treatment is the standard today for treating children with MAM.
  Arms: Current protocol

SUMMARY:
The long-term objective of this proposal is to develop and demonstrate an effective, integrated and streamlined protocol to treat moderate acute malnutrition (MAM) and non-complicated severe acute malnutrition (SAM) in children during humanitarian emergencies.

Hypothesis: An integrated management protocol for MAM and SAM will achieve greater community coverage and a greater individual recovery rate than standard care.

DETAILED DESCRIPTION:
Specific Aim 1: Implement an integrated protocol in Sierra Leone for the management of MAM and non-complicated SAM that uses a single anthropometric indicator as well as the same food. Standard care refers to traditional, segregated treatment of MAM and SAM.

Hypothesis: An integrated management protocol for MAM and SAM will achieve greater community coverage and a greater individual recovery rate than standard care.

Methods Eligible subjects will be children with MAM or non-complicated SAM aged 6-59 months. MAM is defined as MUAC < 12.5 cm, but ≥ 11.5 cm. Non-complicated SAM will be defined as MUAC < 11.5 cm, or + or ++ bilateral edema, and having an acceptable appetite. An acceptable appetite will be judged by giving the child 30 g of RUTF and asking the mother to feed this food to the child over 20 minutes. Children with SAM who are able to consume this RUTF will be eligible for the study. Children unable to consume the RUTF or presenting with IMCI warning signs (convulsions, altered mental status, respiratory distress) will be considered to have complicated SAM and will be referred for inpatient treatment. Only the youngest child with malnutrition in each household will be enrolled; older siblings will be treated operationally using the same protocol. Exclusion criteria include children with obvious chronic debilitating illness like cerebral palsy or congenital abnormalities, or having received treatment for MAM or SAM in the previous two months. If any child needs immediate medical care s/he will be offered treatment or transport to the nearest health center, and not enrolled.

Informed consent will be sought from the caretakers of all eligible children by a nurse familiar with the study and fluent in the caretaker's native language. Duration of the study and participation requirements will be explained. Informed consent will be given verbally and in writing.

Study design This is a cluster randomized, unblinded, clinical controlled trial conducted in children comparing integrated treatment of SAM and MAM with standard treatment. The primary outcomes will be treatment coverage and recovery rate. The very obvious differences in integrated and standard care makes subject and staff blinding impossible.

Ten study sites in rural and peri-urban Sierra Leone, where treatment for SAM and MAM is currently offered, will be selected by the Ministry of Health and Sanitation National Nutrition Program Sierra Leone and the PI for the study. Site managers will be consulted and their cooperation will be solicited prior to definitively selecting sites.

The minimum sample size will be 900 children with MAM and 900 with SAM, 450 receiving integrated care and 450 receiving standard care in each group. Assuming that recovery rate is 75%, this sample size will detect an improvement in the recovery rate to 80% on the integrated protocol, with 95% specificity and 82% power.

Participation Integrated Protocol Upon enrollment demographic information will be collected, weight, height and MUAC will be measured, simple health history obtained, and children will be assessed for edema. Information will be recorded on a standard data collection card. Enough RUTF will be dispensed for 2 weeks of therapy, and children will be asked to return for follow-up every 2 weeks. Children with SAM will initially be given oral amoxicillin twice daily for a week and asked to return for follow-up every 2 weeks. Once children with SAM achieve MUAC >11.5 cm, the RUTF dose will be reduced.

Upon follow-up, caretakers of children will be questioned about symptoms of acute illness, compliance with study foods and food intolerance or allergy. If edema persists or MUAC is ≤ 12.5 cm, an additional two weeks of RUTF will be dispensed. If the child is judged to have altered mental status, respiratory distress or an acute clinical illness needing medical care, the child will be referred to the health center for complicated SAM and withdrawn.

If MUAC > 12.5 cm, the child will be given lipid-based nutrient supplements (LNS), a bed net, albendazole, zinc, referral for immunizations compliant with current WHO recommendations, oral rehydration salts to give if the child has more than three loose watery stools in 24 hours, and asked to return for follow-up in 1, 3 and 6 months. Caretakers will be instructed to seek medical care sooner if the child has fever, poor appetite or signs of an acute illness.

If the child is between 6-24 months of age, the caretaker will participate in enhanced breastfeeding counseling, carried out by the Care Group model. A Care Group is a team of 10 to 15 trained volunteers who provide health and nutrition education to residents within 10 to 15 households each, with the aim of changing behavior and health practices. Each integrated program center will implement one or several Care Groups depending on the number of 6-24 month old children enrolled in the program. The Care Group model is built upon multiplication of volunteer effort, peer support and community mobilization, thereby creating a social movement involving the entire community to foster positive behavior change. The key message is appropriate complementary feeding with continued breastfeeding in 6-24 month old children. Ancillary messages to be included are family planning, immediate and exclusive breastfeeding of infants 0-5 months, and safe hygiene practices. All health and community health workers involved in the project will follow a one week Care Group training to support adequate complementary feeding for the 6-24 month olds.

Participation Standard Protocol These children will receive treatment in accordance with the 'National protocol for community-based management of acute malnutrition' of Sierra Leone, which reflects standard practice worldwide. The management scheme uses weight-for-height z-score (WHZ) to categorize children and includes separate care for MAM and non-complicated SAM, using different foods.

A research assistant will be assigned to the standard care sites to collect informed consent, data, and to assess the availability of foods and supplies. If food is not available, the study will supply, as it is essential for making a valid comparison between the two protocols.

Integrated Protocol Foods Children participating in the integrated treatment protocol will receive, as a supplement to the normal diet, 75 kcal/kg/d RUTF when MUAC ≥ 11.5 cm and edema has resolved, whether s/he was enrolled for MAM or SAM. Children with MUAC < 11.5 cm will receive 175 kcal/kg/d RUTF. Caretakers will be instructed to give her child the appropriate food for the child's nutritional status.

RUTF for the integrated program will be formulated to comply with the new United Nations (UN) ready-to-use supplemental food (RUSF) requirements. RUTF for a 7.5 kg child at 75 kcal/kg/d meets or exceeds the Dietary Reference Intake, except for calcium, phosphorus, potassium, riboflavin and vitamin K, which should be provided in breast milk or the habitual diet.

Children randomized to be in the integrated protocol group will be given a six-week supply of a 50 g LNS to complement their home diet after graduation. LNS is a mixture of peanut butter, fat and the correct mixture of micronutrients to achieve one Required Daily Amounts (RDA)/d for most vitamins and minerals.

Coverage The Simplified Lot Quality Assurance Sampling (LQAS) Evaluation of Access and Coverage (SLEAC) method will be used to assess coverage. The ten treatment centers (five standard and five integrated) will each be assessed for coverage using simple surveys. SLEAC identifies the category of coverage (e.g. low, medium, high) of each treatment center, according to a threshold value, d, calculated as follows: where n is the sample size and p is the standard against which coverage is being evaluated. The Sphere minimum standard of coverage is 50% for rural areas, 70% for urban areas and 90% for camp settings11, so p = 50% for coverage assessments in rural areas, and d = 21 in this scenario. The sample size for each treatment center, n, is 42 (single sided test, 90% power, 5% significance with a control coverage estimated at 20% and intervention coverage estimated at 50%). Since it is likely that more than the exact number of cases will be found, d will be recalculated after coverage assessment. Villages to be visited for surveying are determined by the centric systematic area sampling or quadrat method (selects villages to visit based on geographic location), or by listing all villages and systematically selecting villages in the targeted catchment area for the program, depending on whether a map is available. Sampling ceases after all selected villages are visited, regardless of whether the quota of cases is achieved earlier or not.

House-to-house sampling must be carried out to ensure that all MAM cases are found. This will additionally allow discovery of all SAM cases. Surveying of 14 areas with 15 mid-level health management staff and one principal surveyor required 44 days. It will take the same staff size ~32 working days to complete the survey for this protocol.

Data Analysis Anthropometric indices will be calculated using Anthro v 3.1 (WHO) based on the WHO's 2006 Child Growth Standards. Data will be tabulated and analyzed using the statistical computer program SPSS 13.0 and Microsoft® Excel. A primary outcome is recovery under the integrated program and the standard protocol. Recovery at 1, 3 and 6 months follow-up with the standard protocol will be compared to the integrated protocol. The other primary outcome, coverage, is assessed by comparing survey data from each region; the number of cases found that have been treated are compared to the threshold value, d, and areas are categorized as having low, moderate or high coverage. All coverage analysis will be carried out according to previous published methods.

Secondary outcomes are growth rates, duration of treatment, cost estimates for participation, reasons for defaulting and identification of risk factors for poor outcomes. Comparisons between treatments will be made using Chi-square test for categorical outcomes and ANOVA for continuous outcomes. P < 0.05 will be statistically significant.

Specific Aim 2 will be conducted by International Medical Corps (IMC) Specific Aim 2: Evaluate the effectiveness of breastfeeding education and counseling on breast milk intake in 6-24 month-old children receiving RUTF in Sierra Leone.

Hypothesis: An active, peer counseling program to preserve/promote breastfeeding in MAM infants will result in greater breast milk consumption than standard care.

Methods Subjects: Eligible subjects will be children aged 6-24 months enrolled in the trial described in Specific Aim 1 that have reached MUAC > 12.5 cm. IMC will enroll children between 6-24 months of age whose caretaker will participate in enhanced breastfeeding counseling, carried out by the Care Group model or a modified version tailored to the context of the research program.

Study design IMC will assist each integrated program center to implement one or several Care Groups depending on the number of 6-24 month old children enrolled in the program. The key message for this group of care givers will focus on appropriate complementary feeding with continued breastfeeding in 6-24 month old children Ancillary messages to be included are family planning, health care seeking behaviors, and safe hygiene practices. IMC will train all community health workers involved in the project in a one week intensive training on the Care Group approach to support adequate complementary feeding for the 6-24 month olds.

Participation Caretakers will be approached for sub study enrollment immediately upon successful completion of therapy for MAM, during the interval when their children are receiving the LNS.

It is anticipated that the children whose mother received the Care Group counseling will have greater breast milk intake. There are ample numbers of eligible children in the study such that if a mother chooses not to participate or drops out after agreeing, a replacement can be easily found.

ELIGIBILITY:
Inclusion Criteria:

* Children with MAM or non-complicated SAM aged 6-59 months.
* Have an acceptable appetite.judged by giving the child 30 g of RUTF and asking the mother to feed this food to the child over 20 minutes. Children with SAM who are able to consume this RUTF will be eligible for the study. Children unable to consume the RUTF or presenting with IMCI warning signs (convulsions, altered mental status, respiratory distress) will be considered to have complicated SAM and will be referred for inpatient treatment.
* Only the youngest child with malnutrition in each household will be enrolled; older siblings with MAM or SAM will be treated operationally using the same protocol.

Exclusion Criteria:

* Children with obvious chronic debilitating illness like cerebral palsy or congenital abnormalities
* Children having received treatment for MAM or SAM in the previous two months.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1957 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Project Peanut Butter Factory - 41D Wilkinson Road, Freetown, Sierra Leone

REFERENCES:
- [Background] Myatt M, Khara T, Collins S. A review of methods to detect cases of severely malnourished children in the community for their admission into community-based therapeutic care programs. Food Nutr Bull. 2006 Sep;27(3 Suppl):S7-23. doi: 10.1177/15648265060273S302. PMID 17076211
- [Background] Islam MM, Khatun M, Peerson JM, Ahmed T, Mollah MA, Dewey KG, Brown KH. Effects of energy density and feeding frequency of complementary foods on total daily energy intakes and consumption of breast milk by healthy breastfed Bangladeshi children. Am J Clin Nutr. 2008 Jul;88(1):84-94. doi: 10.1093/ajcn/88.1.84. PMID 18614728
- [Background] Nackers F, Broillet F, Oumarou D, Djibo A, Gaboulaud V, Guerin PJ, Rusch B, Grais RF, Captier V. Effectiveness of ready-to-use therapeutic food compared to a corn/soy-blend-based pre-mix for the treatment of childhood moderate acute malnutrition in Niger. J Trop Pediatr. 2010 Dec;56(6):407-13. doi: 10.1093/tropej/fmq019. Epub 2010 Mar 23. PMID 20332221
- [Background] LaGrone LN, Trehan I, Meuli GJ, Wang RJ, Thakwalakwa C, Maleta K, Manary MJ. A novel fortified blended flour, corn-soy blend "plus-plus," is not inferior to lipid-based ready-to-use supplementary foods for the treatment of moderate acute malnutrition in Malawian children. Am J Clin Nutr. 2012 Jan;95(1):212-9. doi: 10.3945/ajcn.111.022525. Epub 2011 Dec 14. PMID 22170366
- [Background] Oakley E, Reinking J, Sandige H, Trehan I, Kennedy G, Maleta K, Manary M. A ready-to-use therapeutic food containing 10% milk is less effective than one with 25% milk in the treatment of severely malnourished children. J Nutr. 2010 Dec;140(12):2248-52. doi: 10.3945/jn.110.123828. Epub 2010 Oct 27. PMID 20980648
- [Background] Galpin L, Thakwalakwa C, Phuka J, Ashorn P, Maleta K, Wong WW, Manary MJ. Breast milk intake is not reduced more by the introduction of energy dense complementary food than by typical infant porridge. J Nutr. 2007 Jul;137(7):1828-33. doi: 10.1093/jn/137.7.1828. PMID 17585038
- [Result] Maust A, Koroma AS, Abla C, Molokwu N, Ryan KN, Singh L, Manary MJ. Severe and Moderate Acute Malnutrition Can Be Successfully Managed with an Integrated Protocol in Sierra Leone. J Nutr. 2015 Nov;145(11):2604-9. doi: 10.3945/jn.115.214957. Epub 2015 Sep 30. PMID 26423737
- See also: WHO Multicentre Growth Reference Study Group. WHO Child Growth Standards: Length/ height-for-age, weight-for-age, weight-for-length, weight-for-height and body mass index-for-age: Methods and development. Geneva; 2006 — http://www.ncbi.nlm.nih.gov/pubmed/22251429.
- See also: Measuring the effectiveness of Supplementary Feeding Programmes in emergencies. Humanitarian Practice Network. 2008 — https://odihpn.org/resources/measuring-the-effectiveness-of-supplementary-feeding-programmes-in-emergencies/
- See also: World Relief. The Care Group Difference — http://coregroup.secure.nonprofitsoapbox.com/our-technical-work/working-groups/nutrition
- See also: Anon. The U.S. President's Emergency Plan for AIDS Relief — http://www.pepfar.gov/documents/organization/133035.pdf
- See also: World Health Organization and UNICEF. Integrated Management of Childhood Illness (IMCI) Handbook. Geneva; 2005 — http://whqlibdoc.who.int/publications/2005/9241546441.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Integrated Protocol: Integrated protocol for treatment of children with MAM and SAM in humanitarian emergencies has the potential to result in a more streamlined, cost-effective program, higher recovery, and higher program coverage, allowing easier access to malnourished children, thus curing more children of malnutrition and preventing its lifelong effects.
  Integrated Protocol: Implement an integrated protocol in Sierra Leone for the management of MAM and non-complicated SAM that uses a single anthropometric indicator as well as the same food but in different doses to treat the continuum of malnutrition. MAM children will be given 75 g/kg/day of RUTF whereas SAM will be given 175 gr/kg/day of RUTF until MUAC>12.5 cm is reached. Then child will be given LNS, a bed net, albendazole, zinc, referral for immunizations compliant with current WHO recommendations, oral rehydration salts to give if the child has more than three loose watery stools in 24 hours, and asked to return for follow-up in 1, 3 and 6 m
Period: Overall Study
Arm/Group | Integrated Protocol | Current Protocol
Started | 1100 | 857
Completed | 1100 | 857
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Protocol | Current Protocol | Total
Number analyzed (Participants) | 1100 | 857 | 1957
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.7 (8.6) | 14.5 (7.8) | 14.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 619 | 478 | 1097
  Male | 481 | 379 | 860
Region of Enrollment [Number; unit: participants]
  Sierra Leone | 1100 | 857 | 1957
Midupper arm circumference [Mean (Standard Deviation); unit: cm] | 12.1 (0.3) | 11.4 (1.0) | 11.8 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Recovery Under the Integrated Program and the Standard Protocol
Description: Recovery by the end of treatment standard protocol will be compared to the integrated protocol. Recovery will be defined as mid upper arm circumference (MUAC) reaching ≥12.5 cm.
  Subjects will return to clinic every 2 weeks until MUAC of 12.5 cm is reached or until 12 weeks has elapsed.
Time Frame: 12 weeks
Population: Recovery was defined as mid upper arm circumference ≥12.5 cm.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Protocol | Current Protocol
Number analyzed (Participants) | 1100 | 857
Participants | 910 | 682

2. Secondary Outcome: Change in Growth Rates
Description: Subjects will return to clinic every 2 weeks until MUAC of 12.5 cm is reached or until 12 weeks has elapsed. Measurement is taken at each visit but final recovery measurement will be used.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Integrated Protocol | Current Protocol
Number analyzed (Participants) | 1100 | 857
cm | 0.52 (0.04) | 0.25 (0.02)

3. Secondary Outcome: Duration of Treatment
Description: Subjects will return to clinic every 2 weeks until MUAC of 12.5 cm is reached or until 12 weeks has elapsed. Time to achieve MUAC of 12.5 cm will be documented.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Number of clinic visits
Arm/Group | Integrated Protocol | Current Protocol
Number analyzed (Participants) | 1100 | 857
Number of clinic visits | 2.7 (0.06) | 3.5 (0.07)

4. Secondary Outcome: Change in Recovery Status After 12 Weeks
Description: Any changes in recovery will be measured 6 months at follow-up visit. Number of children still well nourished.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated Protocol | Current Protocol
Number analyzed (Participants) | 604 | 474
Participants | 544 | 459

ADVERSE EVENTS:
Arm/Group | Integrated Protocol | Current Protocol
All-Cause Mortality (participants affected / at risk) | 42/1100 | 35/857
Serious Adverse Events (participants affected / at risk) | 0/1100 | 0/857
Other Adverse Events (participants affected / at risk) | 0/1100 | 0/857

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No